CLINICAL TRIAL: NCT05225025
Title: A Pilot Trial of the ROSE Postpartum Depression Prevention Intervention in Antepartum Patients Admitted to High-risk Obstetrics Unit
Brief Title: A Pilot Trial of the Reach Out, Stay Strong, Essentials for Mothers of Newborns (ROSE) Postpartum Depression Prevention Intervention in Pregnant Patients Admitted to Strong Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Mae Stone Goode Foundation (Other)
Responsible Party: Principal Investigator, Ellen Poleshuck, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005941
Record Dates: First submitted 2022-01-07; First posted 2022-02-04 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Depression; Postpartum Anxiety
MeSH Terms: conditions — Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSE Intervention (Experimental)
  Interventions: Behavioral: ROSE
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: ROSE — The ROSE (Reach Out, Stay Strong, Essentials for mothers of newborns) program is an evidence-based intervention that has been proven to reduce cases of post-partum depression among low-income and racially and ethnically diverse women.
  ROSE is administered to pregnant women in small group settings, typically in the same location that prenatal care is being provided (in this study, a hospital setting). It is divided into four 90-minute group sessions and teaches interpersonal psychotherapy-based skills that mitigate identified risk factors for PPD such as social support, stress management skills and communication.
  ROSE curriculum will be implemented using groups in a continuous cycle, with patients entering into the intervention curriculum at the time of their enrollment and continuing through until all 4 total sessions have been accomplished.
  Arms: ROSE Intervention
Other: Standard of Care — Usual hospital care with no behavioral intervention
  Arms: Standard of Care

SUMMARY:
This study is a pilot, single-center, randomized controlled trial. It will

1. determine feasibility and acceptability of an evidence-based intervention for prevention of postpartum depression with antepartum patients on a high-risk obstetric unit,
2. determine what adaptations may be needed for an inpatient population
3. determine what retention strategies are most successful and acceptable for this patient population
4. estimate the effect size of an intervention for in-hospital distress, anxiety and depression
5. estimate the effect size of an intervention to reduce the risk of a post-partum depression diagnosis or depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Viable pregnancy between 20 weeks 0 days and 35 weeks 0 days gestation at the time of enrollment
* Anticipated admission to the hospital for >5 days due to pregnancy complication requiring hospital observation
* Age > 18 years
* Planned hospitalization at Strong Memorial Hospital through the duration of antepartum course
* Planned delivery at Strong Memorial Hospital

Exclusion Criteria:

* Fetal demise in utero
* Inability to give informed consent secondary to intellectual capacity
* English is not primary language used to communicate
* Currently incarcerated
* Age < 18 years
* Planned antepartum hospitalization at another institution
* Planned delivery at another institution
* Actively suicidal or in need of acute psychiatric care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Subject-reported in-hospital distress | 14 days
  Hospital distress will be measured using the Depression, Anxiety and Stress Scale-21 (DASS-21) Stress subscale. Stress subscale ranges from 0 to 42 with higher scores indicating worse outcome.
Subject-reported depressive symptom severity | 6 weeks postpartum
  Depressive symptom severity will be measured using the Edinburgh Postnatal Depression Scale (EPDS). The scale ranges from 0-30 with higher scores indicating worse outcome.
Subject-reported anxiety symptom severity | 6 weeks postpartum
  Anxiety symptom severity will be measured using the General Anxiety Disorder-7 (GAD-7) measurement scale. The scale ranges from 0 to 21 with higher scores indicating worse outcome.
Clinical diagnosis of depression | 6 weeks postpartum
  Diagnosis of depression will be made using the Mini International Neuropsychiatric Interview (M.I.N.I) brief structured diagnostic interview which explores, in a standardized way, the main psychiatric disorders of Axis I of the DSM-IV TR. Only modules A and B (Major depressive episode and dysthymia) will be used. This structured interview contains questions with binary answers, with Yes indicating worse outcome.

OTHER OUTCOMES:
satisfaction with ROSE behavioral health intervention | 14 days and 6 weeks postpartum
  Satisfaction score will be measured using the Client Satisfaction Questionnaire-8 (CSQ-8). The scores range from 8-32, with greater satisfaction indicated by higher scores.
self-reported mother-infant bonding | 6 weeks postpartum
  Mother-infant bonding will be assessed over four domains by the Postpartum Bonding Questionnaire (PBQ). Scores range from 0-125, with worse outcome indicated by higher scores.
self-reported functional status | 6 weeks postpartum
  Functional status will be assessed using the Inventory of Functional Status After Childbirth (IFSAC) measure. Scores range from 36-144, with higher scores indicating better outcome.
percentage of eligible subjects who enrolled in the study | baseline
percentage of enrolled subjects who completed all inpatient study activities | 14 days
percentage of enrolled subjects who completed all inpatient plus outpatient study activities | 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Strong Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No